CLINICAL TRIAL: NCT02591615
Title: Randomized Phase II Trial Evaluating the Optimal Sequencing of PD-1 Inhibition With Pembrolizumab (MK-3475) and Standard Platinum-based Chemotherapy in Patients With Chemotherapy Naive Stage IV Non-small Cell Lung Cancer
Brief Title: Optimal Sequencing of Pembrolizumab (MK-3475) and Standard Platinum-based Chemotherapy in First-Line NSCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance Foundation Trials, LLC. (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AFT-09
Record Dates: First submitted 2015-10-20; First posted 2015-10-29 (Estimated); Results first posted 2022-12-28 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-11

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab; Carboplatin; Paclitaxel; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Active Comparator): For Squamous Carcinoma Carboplatin AUC = 6 IV day 1 every 21-days for up to 4 cycles Paclitaxel 200 mg/m2 IV day 1 every 21-days for up to 4 cycles
  OR
  For Non-squamous Carcinoma Carboplatin AUC = 6 IV day 1 every 21-days for up to 4 cycles Pemetrexed 500 mg/m2 IV day 1 every 21-days for up to 4 cycles
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Drug: Pemetrexed
- Arm B (Active Comparator): MK-3475 200 mg/m2 IV every 21-days for up to 4 cycles
  Patients with CR, PR, or SD by irRC will then be treated with:
  For Squamous Carcinoma:
  Carboplatin AUC = 6 IV day 1 every 21-days for up to 4 cycles Paclitaxel 200 mg/m2 IV day 1 every 21-days for up to 4 cycles
  OR
  For Non-squamous Carcinoma
  Carboplatin AUC = 6 IV day 1 every 21-days for up to 4 cycles Pemetrexed 500 mg/m2 IV day 1 every 21-days for up to 4 cycles
  Interventions: Drug: MK-3475; Drug: Carboplatin; Drug: Paclitaxel; Drug: Pemetrexed

INTERVENTIONS:
Drug: MK-3475 — Dose frequency of Q3W, Day 1 of each cycle
  Other Names: Pembrolizumab
  Arms: Arm B
Drug: Carboplatin — Dose frequency of Q3W, Day 1 of each cycle (standard Chemotherapy)
  Other Names: Paraplat; Paraplatin
Drug: Paclitaxel — Dose frequency of Q3W, Day 1 of each cycle (standard Chemotherapy)
  Other Names: Taxol
Drug: Pemetrexed — Dose frequency of Q3W, Day 1 of each cycle (standard Chemotherapy)
  Other Names: Alimta

SUMMARY:
This is a multicenter randomized phase II to determine if the administration of standard platinum-based chemotherapy before MK-3475 in with Chemotherapy naive stage IV Non-small Cell Lung Cancer (NSCLC) will improve the overall response rate (ORR) compared to MK-3475 administered before chemotherapy. Patients will be given Pembrolizumab as maintenance up to 2 years: Carboplatin and paclitaxel or pemetrexed every 3 weeks x 4 cycles followed by pembrolizumab every 3 weeks for up to 2 years. Pembrolizumab every 3 weeks x 4 cycles followed by carboplatin and paclitaxel or pemetrexed every 3 weeks x 4 cycles followed by pembrolizumab every 3 weeks for up to 2 years.

DETAILED DESCRIPTION:
While a genotype-directed strategy has been established as effective in treatment selection for patients with advanced NSCLC, only a minority of patients at this time will have a readily identifiable actionable molecular target. Furthermore, genotype-directed therapy has not been validated for patients with squamous cell carcinoma of the lung. Therefore, the majority of patients with advanced NSCLC will continue to rely on standard platinum-based doublet chemotherapy. Given the plateau in effectiveness of this approach, novel treatment strategies are clearly warranted.

ELIGIBILITY:
Inclusion Criteria:

1. Be ≥ 18 years of age on day of signing informed consent.
2. Have a life expectancy of at least 3 months.
3. Have a histologically or cytologically confirmed diagnosis of stage IV NSCLC.
4. Have a performance status of 0 or 1 on the ECOG.
5. Have a measurable disease based on RECIST 1.1.
6. Have provided tissue from an archival tissue sample or newly obtained core or excisional biopsy of tumor lesion.
7. In patients with non-squamous non-small cell lung cancer, investigators must be able to produce source documentation of the EGFR mutation status or ALK translocation status.
8. Demonstrate adequate organ function.
9. Female patient of childbearing potential should have a negative urine or serum pregnancy test within 72 hours.
10. Female parents of childbearing potential must be willing to use 2 methods of birth control or be surgically sterile.
11. Male patients must agree to use an adequate method of contraception.
12. Patients with sensitizing EGFR mutation or ALK rearrangement must have progressed on an appropriate tyrosine kinase inhibitor (TKI)

Exclusion Criteria:

1. Has received prior treatment with chemotherapy or biologic therapy for stage IV NSCLC.
2. Is currently participating in or has participated in a study of an investigational agent or using an investigational device.
3. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy.
4. Has had a prior mAb within 4 weeks prior to study Day 1 or who has not recovered from adverse events due to agents administered more than 4 weeks earlier.
5. Has had prior chemotherapy or radiation.
6. Has a known additional malignancy that is progressing or requires active treatment.
7. Has known active CNS metastases and/or carcinomatous meningitis.
8. Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents.
9. Has evidence of interstitial lung disease or active, non-infectious pneumonitis.
10. Has an active infection requiring systemic therapy.
11. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial.
12. Has known psychiatric or substance abuse disorders.
13. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial.
14. Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or CTLA-4 antibody.
15. Has a known history of HIV.
16. Has known active Hepatitis B or Hepatitis C.
17. Has received a live vaccine within 30 days prior to the planned first dose of study therapy.
18. Has a known history of active TB.
19. Hypersensitivity to pembrolizumab or any of it's excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2019-01-04 (Actual); Study Completion 2020-07-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Monica Bertagnolli, MD, Principal Investigator — Alliance Foundation Trials, LLC.; Thomas Hensing, MD, Study Chair — Endeavor Health
Locations (11):
- United States (11):
  - UCSD Moores Cancer Center, La Jolla, California
  - The University of Chicago Medical Center, Chicago, Illinois
  - NorthShore University HealthSystem, Evanston, Illinois
  - Medical Oncology & Hematology Associates, Des Moines, Iowa
  - EMMC Cancer Care, Brewer, Maine
  - Metro MN Community Oncology Research Consortium, Minneapolis, Minnesota
  - NH Oncology (Concord), Concord, New Hampshire
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - SUNY Upstate Medical University, Syracuse, New York
  - The Ohio State University, Columbus, Ohio
  - University of Oklahoma Health Sciences Center Stephenson Cancer Center, Oklahoma City, Oklahoma

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Siegel R, Ma J, Zou Z, Jemal A. Cancer statistics, 2014. CA Cancer J Clin. 2014 Jan-Feb;64(1):9-29. doi: 10.3322/caac.21208. Epub 2014 Jan 7. PMID 24399786
- [Background] Socinski MA, Evans T, Gettinger S, Hensing TA, VanDam Sequist L, Ireland B, Stinchcombe TE. Treatment of stage IV non-small cell lung cancer: Diagnosis and management of lung cancer, 3rd ed: American College of Chest Physicians evidence-based clinical practice guidelines. Chest. 2013 May;143(5 Suppl):e341S-e368S. doi: 10.1378/chest.12-2361. PMID 23649446
- [Background] Schiller JH, Harrington D, Belani CP, Langer C, Sandler A, Krook J, Zhu J, Johnson DH; Eastern Cooperative Oncology Group. Comparison of four chemotherapy regimens for advanced non-small-cell lung cancer. N Engl J Med. 2002 Jan 10;346(2):92-8. doi: 10.1056/NEJMoa011954. PMID 11784875
- [Background] Sandler A, Gray R, Perry MC, Brahmer J, Schiller JH, Dowlati A, Lilenbaum R, Johnson DH. Paclitaxel-carboplatin alone or with bevacizumab for non-small-cell lung cancer. N Engl J Med. 2006 Dec 14;355(24):2542-50. doi: 10.1056/NEJMoa061884. PMID 17167137
- [Background] Johnson DH, Fehrenbacher L, Novotny WF, Herbst RS, Nemunaitis JJ, Jablons DM, Langer CJ, DeVore RF 3rd, Gaudreault J, Damico LA, Holmgren E, Kabbinavar F. Randomized phase II trial comparing bevacizumab plus carboplatin and paclitaxel with carboplatin and paclitaxel alone in previously untreated locally advanced or metastatic non-small-cell lung cancer. J Clin Oncol. 2004 Jun 1;22(11):2184-91. doi: 10.1200/JCO.2004.11.022. PMID 15169807
- [Background] Scagliotti GV, Parikh P, von Pawel J, Biesma B, Vansteenkiste J, Manegold C, Serwatowski P, Gatzemeier U, Digumarti R, Zukin M, Lee JS, Mellemgaard A, Park K, Patil S, Rolski J, Goksel T, de Marinis F, Simms L, Sugarman KP, Gandara D. Phase III study comparing cisplatin plus gemcitabine with cisplatin plus pemetrexed in chemotherapy-naive patients with advanced-stage non-small-cell lung cancer. J Clin Oncol. 2008 Jul 20;26(21):3543-51. doi: 10.1200/JCO.2007.15.0375. Epub 2008 May 27. PMID 18506025
- [Background] Scagliotti G, Brodowicz T, Shepherd FA, Zielinski C, Vansteenkiste J, Manegold C, Simms L, Fossella F, Sugarman K, Belani CP. Treatment-by-histology interaction analyses in three phase III trials show superiority of pemetrexed in nonsquamous non-small cell lung cancer. J Thorac Oncol. 2011 Jan;6(1):64-70. doi: 10.1097/JTO.0b013e3181f7c6d4. PMID 21119545
- [Background] Mok TS, Wu YL, Thongprasert S, Yang CH, Chu DT, Saijo N, Sunpaweravong P, Han B, Margono B, Ichinose Y, Nishiwaki Y, Ohe Y, Yang JJ, Chewaskulyong B, Jiang H, Duffield EL, Watkins CL, Armour AA, Fukuoka M. Gefitinib or carboplatin-paclitaxel in pulmonary adenocarcinoma. N Engl J Med. 2009 Sep 3;361(10):947-57. doi: 10.1056/NEJMoa0810699. Epub 2009 Aug 19. PMID 19692680
- [Background] Maemondo M, Inoue A, Kobayashi K, Sugawara S, Oizumi S, Isobe H, Gemma A, Harada M, Yoshizawa H, Kinoshita I, Fujita Y, Okinaga S, Hirano H, Yoshimori K, Harada T, Ogura T, Ando M, Miyazawa H, Tanaka T, Saijo Y, Hagiwara K, Morita S, Nukiwa T; North-East Japan Study Group. Gefitinib or chemotherapy for non-small-cell lung cancer with mutated EGFR. N Engl J Med. 2010 Jun 24;362(25):2380-8. doi: 10.1056/NEJMoa0909530. PMID 20573926
- [Background] Mitsudomi T, Morita S, Yatabe Y, Negoro S, Okamoto I, Tsurutani J, Seto T, Satouchi M, Tada H, Hirashima T, Asami K, Katakami N, Takada M, Yoshioka H, Shibata K, Kudoh S, Shimizu E, Saito H, Toyooka S, Nakagawa K, Fukuoka M; West Japan Oncology Group. Gefitinib versus cisplatin plus docetaxel in patients with non-small-cell lung cancer harbouring mutations of the epidermal growth factor receptor (WJTOG3405): an open label, randomised phase 3 trial. Lancet Oncol. 2010 Feb;11(2):121-8. doi: 10.1016/S1470-2045(09)70364-X. Epub 2009 Dec 18. PMID 20022809
- [Background] Zhou C, Wu YL, Chen G, Feng J, Liu XQ, Wang C, Zhang S, Wang J, Zhou S, Ren S, Lu S, Zhang L, Hu C, Hu C, Luo Y, Chen L, Ye M, Huang J, Zhi X, Zhang Y, Xiu Q, Ma J, Zhang L, You C. Erlotinib versus chemotherapy as first-line treatment for patients with advanced EGFR mutation-positive non-small-cell lung cancer (OPTIMAL, CTONG-0802): a multicentre, open-label, randomised, phase 3 study. Lancet Oncol. 2011 Aug;12(8):735-42. doi: 10.1016/S1470-2045(11)70184-X. Epub 2011 Jul 23. PMID 21783417
- [Background] Rosell R, Carcereny E, Gervais R, Vergnenegre A, Massuti B, Felip E, Palmero R, Garcia-Gomez R, Pallares C, Sanchez JM, Porta R, Cobo M, Garrido P, Longo F, Moran T, Insa A, De Marinis F, Corre R, Bover I, Illiano A, Dansin E, de Castro J, Milella M, Reguart N, Altavilla G, Jimenez U, Provencio M, Moreno MA, Terrasa J, Munoz-Langa J, Valdivia J, Isla D, Domine M, Molinier O, Mazieres J, Baize N, Garcia-Campelo R, Robinet G, Rodriguez-Abreu D, Lopez-Vivanco G, Gebbia V, Ferrera-Delgado L, Bombaron P, Bernabe R, Bearz A, Artal A, Cortesi E, Rolfo C, Sanchez-Ronco M, Drozdowskyj A, Queralt C, de Aguirre I, Ramirez JL, Sanchez JJ, Molina MA, Taron M, Paz-Ares L; Spanish Lung Cancer Group in collaboration with Groupe Francais de Pneumo-Cancerologie and Associazione Italiana Oncologia Toracica. Erlotinib versus standard chemotherapy as first-line treatment for European patients with advanced EGFR mutation-positive non-small-cell lung cancer (EURTAC): a multicentre, open-label, randomised phase 3 trial. Lancet Oncol. 2012 Mar;13(3):239-46. doi: 10.1016/S1470-2045(11)70393-X. Epub 2012 Jan 26. PMID 22285168
- [Background] Yang, J.C., et al., Overall Survival in Patients with Advanced Non-small Cell Lung Cancer Harboring Common (Del 19/L858R) Epidermal Growth Factor Receptor Mutations: Pooled Analysis of Two Large Open-label Phase III Studies Comparing Afatinib with Chemotherapy. J Clin Oncol, 2014. 32:5s((suppl; abstr 8004))
- [Background] Shaw AT, Kim DW, Nakagawa K, Seto T, Crino L, Ahn MJ, De Pas T, Besse B, Solomon BJ, Blackhall F, Wu YL, Thomas M, O'Byrne KJ, Moro-Sibilot D, Camidge DR, Mok T, Hirsh V, Riely GJ, Iyer S, Tassell V, Polli A, Wilner KD, Janne PA. Crizotinib versus chemotherapy in advanced ALK-positive lung cancer. N Engl J Med. 2013 Jun 20;368(25):2385-94. doi: 10.1056/NEJMoa1214886. Epub 2013 Jun 1. PMID 23724913
- [Background] Shaw AT, Kim DW, Mehra R, Tan DS, Felip E, Chow LQ, Camidge DR, Vansteenkiste J, Sharma S, De Pas T, Riely GJ, Solomon BJ, Wolf J, Thomas M, Schuler M, Liu G, Santoro A, Lau YY, Goldwasser M, Boral AL, Engelman JA. Ceritinib in ALK-rearranged non-small-cell lung cancer. N Engl J Med. 2014 Mar 27;370(13):1189-97. doi: 10.1056/NEJMoa1311107. PMID 24670165
- [Background] Disis ML. Immune regulation of cancer. J Clin Oncol. 2010 Oct 10;28(29):4531-8. doi: 10.1200/JCO.2009.27.2146. Epub 2010 Jun 1. PMID 20516428
- [Background] Dong H, Strome SE, Salomao DR, Tamura H, Hirano F, Flies DB, Roche PC, Lu J, Zhu G, Tamada K, Lennon VA, Celis E, Chen L. Tumor-associated B7-H1 promotes T-cell apoptosis: a potential mechanism of immune evasion. Nat Med. 2002 Aug;8(8):793-800. doi: 10.1038/nm730. Epub 2002 Jun 24. PMID 12091876
- [Background] Sharpe AH, Freeman GJ. The B7-CD28 superfamily. Nat Rev Immunol. 2002 Feb;2(2):116-26. doi: 10.1038/nri727. PMID 11910893
- [Background] Brown JA, Dorfman DM, Ma FR, Sullivan EL, Munoz O, Wood CR, Greenfield EA, Freeman GJ. Blockade of programmed death-1 ligands on dendritic cells enhances T cell activation and cytokine production. J Immunol. 2003 Feb 1;170(3):1257-66. doi: 10.4049/jimmunol.170.3.1257. PMID 12538684
- [Background] Francisco LM, Sage PT, Sharpe AH. The PD-1 pathway in tolerance and autoimmunity. Immunol Rev. 2010 Jul;236:219-42. doi: 10.1111/j.1600-065X.2010.00923.x. PMID 20636820
- [Background] Thompson RH, Dong H, Lohse CM, Leibovich BC, Blute ML, Cheville JC, Kwon ED. PD-1 is expressed by tumor-infiltrating immune cells and is associated with poor outcome for patients with renal cell carcinoma. Clin Cancer Res. 2007 Mar 15;13(6):1757-61. doi: 10.1158/1078-0432.CCR-06-2599. PMID 17363529
- [Background] Shepherd FA, Douillard JY, Blumenschein GR Jr. Immunotherapy for non-small cell lung cancer: novel approaches to improve patient outcome. J Thorac Oncol. 2011 Oct;6(10):1763-73. doi: 10.1097/JTO.0b013e31822e28fc. PMID 21876456
- [Background] Hiraoka K, Miyamoto M, Cho Y, Suzuoki M, Oshikiri T, Nakakubo Y, Itoh T, Ohbuchi T, Kondo S, Katoh H. Concurrent infiltration by CD8+ T cells and CD4+ T cells is a favourable prognostic factor in non-small-cell lung carcinoma. Br J Cancer. 2006 Jan 30;94(2):275-80. doi: 10.1038/sj.bjc.6602934. PMID 16421594
- [Background] Zhuang X, Xia X, Wang C, Gao F, Shan N, Zhang L, Zhang L. A high number of CD8+ T cells infiltrated in NSCLC tissues is associated with a favorable prognosis. Appl Immunohistochem Mol Morphol. 2010 Jan;18(1):24-8. doi: 10.1097/PAI.0b013e3181b6a741. PMID 19713832
- [Background] Talmadge JE, Donkor M, Scholar E. Inflammatory cell infiltration of tumors: Jekyll or Hyde. Cancer Metastasis Rev. 2007 Dec;26(3-4):373-400. doi: 10.1007/s10555-007-9072-0. PMID 17717638
- [Background] Usubutun A, Ayhan A, Uygur MC, Ozen H, Toklu C, Ruacan S. Prognostic factors in renal cell carcinoma. J Exp Clin Cancer Res. 1998 Mar;17(1):77-81. PMID 9646237
- [Background] Al-Shibli KI, Donnem T, Al-Saad S, Persson M, Bremnes RM, Busund LT. Prognostic effect of epithelial and stromal lymphocyte infiltration in non-small cell lung cancer. Clin Cancer Res. 2008 Aug 15;14(16):5220-7. doi: 10.1158/1078-0432.CCR-08-0133. PMID 18698040
- [Background] Deschoolmeester V, Baay M, Van Marck E, Weyler J, Vermeulen P, Lardon F, Vermorken JB. Tumor infiltrating lymphocytes: an intriguing player in the survival of colorectal cancer patients. BMC Immunol. 2010 Apr 12;11:19. doi: 10.1186/1471-2172-11-19. PMID 20385003
- [Background] Galon J, Costes A, Sanchez-Cabo F, Kirilovsky A, Mlecnik B, Lagorce-Pages C, Tosolini M, Camus M, Berger A, Wind P, Zinzindohoue F, Bruneval P, Cugnenc PH, Trajanoski Z, Fridman WH, Pages F. Type, density, and location of immune cells within human colorectal tumors predict clinical outcome. Science. 2006 Sep 29;313(5795):1960-4. doi: 10.1126/science.1129139. PMID 17008531
- [Background] Nobili C, Degrate L, Caprotti R, Franciosi C, Leone BE, Trezzi R, Romano F, Uggeri F, Uggeri F. Prolonged survival of a patient affected by pancreatic adenocarcinoma with massive lymphocyte and dendritic cell infiltration after interleukin-2 immunotherapy. Report of a case. Tumori. 2008 May-Jun;94(3):426-30. doi: 10.1177/030089160809400323. PMID 18705415
- [Background] Hodi FS, Dranoff G. The biologic importance of tumor-infiltrating lymphocytes. J Cutan Pathol. 2010 Apr;37 Suppl 1(0 1):48-53. doi: 10.1111/j.1600-0560.2010.01506.x. PMID 20482675
- [Background] Kloor M. Lymphocyte infiltration and prognosis in colorectal cancer. Lancet Oncol. 2009 Sep;10(9):840-1. doi: 10.1016/S1470-2045(09)70245-1. No abstract available. PMID 19717085
- [Background] Lee HE, Chae SW, Lee YJ, Kim MA, Lee HS, Lee BL, Kim WH. Prognostic implications of type and density of tumour-infiltrating lymphocytes in gastric cancer. Br J Cancer. 2008 Nov 18;99(10):1704-11. doi: 10.1038/sj.bjc.6604738. Epub 2008 Oct 21. PMID 18941457
- [Background] Leffers N, Gooden MJ, de Jong RA, Hoogeboom BN, ten Hoor KA, Hollema H, Boezen HM, van der Zee AG, Daemen T, Nijman HW. Prognostic significance of tumor-infiltrating T-lymphocytes in primary and metastatic lesions of advanced stage ovarian cancer. Cancer Immunol Immunother. 2009 Mar;58(3):449-59. doi: 10.1007/s00262-008-0583-5. Epub 2008 Sep 13. PMID 18791714
- [Background] Nishimura H, Honjo T, Minato N. Facilitation of beta selection and modification of positive selection in the thymus of PD-1-deficient mice. J Exp Med. 2000 Mar 6;191(5):891-8. doi: 10.1084/jem.191.5.891. PMID 10704469
- [Background] Hiraoka N. Tumor-infiltrating lymphocytes and hepatocellular carcinoma: molecular biology. Int J Clin Oncol. 2010 Dec;15(6):544-51. doi: 10.1007/s10147-010-0130-1. Epub 2010 Oct 6. PMID 20924634
- [Background] Liotta F, Gacci M, Frosali F, Querci V, Vittori G, Lapini A, Santarlasci V, Serni S, Cosmi L, Maggi L, Angeli R, Mazzinghi B, Romagnani P, Maggi E, Carini M, Romagnani S, Annunziato F. Frequency of regulatory T cells in peripheral blood and in tumour-infiltrating lymphocytes correlates with poor prognosis in renal cell carcinoma. BJU Int. 2011 May;107(9):1500-6. doi: 10.1111/j.1464-410X.2010.09555.x. Epub 2010 Aug 24. PMID 20735382
- [Background] Mu CY, Huang JA, Chen Y, Chen C, Zhang XG. High expression of PD-L1 in lung cancer may contribute to poor prognosis and tumor cells immune escape through suppressing tumor infiltrating dendritic cells maturation. Med Oncol. 2011 Sep;28(3):682-8. doi: 10.1007/s12032-010-9515-2. Epub 2010 Apr 6. PMID 20373055
- [Background] Champiat S, Ileana E, Giaccone G, Besse B, Mountzios G, Eggermont A, Soria JC. Incorporating immune-checkpoint inhibitors into systemic therapy of NSCLC. J Thorac Oncol. 2014 Feb;9(2):144-53. doi: 10.1097/JTO.0000000000000074. PMID 24419410
- [Background] Chen YB, Mu CY, Huang JA. Clinical significance of programmed death-1 ligand-1 expression in patients with non-small cell lung cancer: a 5-year-follow-up study. Tumori. 2012 Nov;98(6):751-5. doi: 10.1177/030089161209800612. PMID 23389362
- [Background] Zhang P, Su DM, Liang M, Fu J. Chemopreventive agents induce programmed death-1-ligand 1 (PD-L1) surface expression in breast cancer cells and promote PD-L1-mediated T cell apoptosis. Mol Immunol. 2008 Mar;45(5):1470-6. doi: 10.1016/j.molimm.2007.08.013. Epub 2007 Oct 24. PMID 17920123
- [Background] Brahmer JR, Tykodi SS, Chow LQ, Hwu WJ, Topalian SL, Hwu P, Drake CG, Camacho LH, Kauh J, Odunsi K, Pitot HC, Hamid O, Bhatia S, Martins R, Eaton K, Chen S, Salay TM, Alaparthy S, Grosso JF, Korman AJ, Parker SM, Agrawal S, Goldberg SM, Pardoll DM, Gupta A, Wigginton JM. Safety and activity of anti-PD-L1 antibody in patients with advanced cancer. N Engl J Med. 2012 Jun 28;366(26):2455-65. doi: 10.1056/NEJMoa1200694. Epub 2012 Jun 2. PMID 22658128
- [Background] Spigel, D., et al., Clinical activity, safety, and biomarkers of MPDL3280A, an engineered PD-L1 antibody in patients with locally advanced or metastic non-small cell lung cancer. J Clin Oncol, 2013. 31(Suppl; abstr 8008).
- [Background] Garon, E., et al., Abstract A20: MK-3475 monotherapy for previously treated non-small cell lung cancer: Preliminary safety and clinical activity. . Clin Cancer Res, 2014. 20: p. A20.
- [Background] Garon, E., et al., Safety and Clinical Activity of MK-3475 in Previously Treated Patients with Non-small Cell Lung CAncer. J Clin Oncol, 2014. 32:5S((suppl;abstr 8020)).
- [Background] Rizvi, N., et al., Safety and Clinical Activity of MK-3475 as Initial Therapy in Patients with Advanced Non-small Cell Lung Cancer. J Clin Oncol, 2014. 32:5s((suppl; abstr 8007)).
- [Background] Gettinger, S.N., et al., First-line Nivolumab Monotherapy in Advanced NSCLC: Safety, Efficacy, and Correlation with PD-L1 Status. . J Clin Oncol, 2014. 325s((suppl; abstr 8024)).
- [Background] Brahmer, J., et al., Survival and long-term follow up of phase I trial of nivolumab (Anti-PD-1; BMS-936558, ONO-4538) in patients with previously treated advanced non-small cell lung cancer. J Clin Oncol, 2013. 31(suppl; abstr 8030).
- [Background] Liu WM, Fowler DW, Smith P, Dalgleish AG. Pre-treatment with chemotherapy can enhance the antigenicity and immunogenicity of tumours by promoting adaptive immune responses. Br J Cancer. 2010 Jan 5;102(1):115-23. doi: 10.1038/sj.bjc.6605465. Epub 2009 Dec 8. PMID 19997099
- [Background] John J, Ismail M, Riley C, Askham J, Morgan R, Melcher A, Pandha H. Differential effects of Paclitaxel on dendritic cell function. BMC Immunol. 2010 Mar 19;11:14. doi: 10.1186/1471-2172-11-14. PMID 20302610
- [Background] Zhang L, Dermawan K, Jin M, Liu R, Zheng H, Xu L, Zhang Y, Cai Y, Chu Y, Xiong S. Differential impairment of regulatory T cells rather than effector T cells by paclitaxel-based chemotherapy. Clin Immunol. 2008 Nov;129(2):219-29. doi: 10.1016/j.clim.2008.07.013. Epub 2008 Sep 3. PMID 18771959
- [Background] Antonia, S.J., et al., Nivolumab (anti-PD-1; BMS-936558, ONO-4538) in combination with platinum-based doublet chemotherapy in advanced non-small cell lung cancer. J Clin Oncol, 2014. 32:5s((suppl; abstr 8113)).
- [Background] Lesterhuis WJ, Salmons J, Nowak AK, Rozali EN, Khong A, Dick IM, Harken JA, Robinson BW, Lake RA. Synergistic effect of CTLA-4 blockade and cancer chemotherapy in the induction of anti-tumor immunity. PLoS One. 2013 Apr 23;8(4):e61895. doi: 10.1371/journal.pone.0061895. Print 2013. PMID 23626745
- [Background] Lynch TJ, Bondarenko I, Luft A, Serwatowski P, Barlesi F, Chacko R, Sebastian M, Neal J, Lu H, Cuillerot JM, Reck M. Ipilimumab in combination with paclitaxel and carboplatin as first-line treatment in stage IIIB/IV non-small-cell lung cancer: results from a randomized, double-blind, multicenter phase II study. J Clin Oncol. 2012 Jun 10;30(17):2046-54. doi: 10.1200/JCO.2011.38.4032. Epub 2012 Apr 30. PMID 22547592
- [Background] Johnson DB, Rioth MJ, Horn L. Immune checkpoint inhibitors in NSCLC. Curr Treat Options Oncol. 2014 Dec;15(4):658-69. doi: 10.1007/s11864-014-0305-5. PMID 25096781
- [Background] Wolchok JD, Hoos A, O'Day S, Weber JS, Hamid O, Lebbe C, Maio M, Binder M, Bohnsack O, Nichol G, Humphrey R, Hodi FS. Guidelines for the evaluation of immune therapy activity in solid tumors: immune-related response criteria. Clin Cancer Res. 2009 Dec 1;15(23):7412-20. doi: 10.1158/1078-0432.CCR-09-1624. Epub 2009 Nov 24. PMID 19934295
- [Background] Simon R, Wittes RE, Ellenberg SS. Randomized phase II clinical trials. Cancer Treat Rep. 1985 Dec;69(12):1375-81. PMID 4075313
- [Background] Fleiss, J., L. B, and M. Paik, Statistical Methods for Rates and Proportions, J.W. Sons, Editor. 2003: New York.

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A Squamous Carcinoma (Platinum Doublet, Then MK-3475, Then Maintenance MK-3475): For Squamous Carcinoma>
  > Carboplatin AUC = 6 IV day 1 every 21-days for up to 4 cycles>
  > Paclitaxel 200 mg/m2 IV day 1 every 21-days for up to 4 cycles>
  >
  >
  > Carboplatin: Dose frequency of Q3W, Day 1 of each cycle (standard Chemotherapy)>
  >
  >
  > Paclitaxel: Dose frequency of Q3W, Day 1 of each cycle (standard Chemotherapy)>
  >
  >
  > Pemetrexed: Dose frequency of Q3W, Day 1 of each cycle (standard Chemotherapy)
- Arm A Non-squamous Carcinoma (Platinum Doublet, Then MK-3475, Then Maintenance MK-3475): For Non-squamous Carcinoma>
  > Carboplatin AUC = 6 IV day 1 every 21-days for up to 4 cycles>
  > Pemetrexed 500 mg/m2 IV day 1 every 21-days for up to 4 cycles>
  > Carboplatin: Dose frequency of Q3W, Day 1 of each cycle (standard Chemotherapy)>
  > Paclitaxel: Dose frequency of Q3W, Day 1 of each cycle (standard Chemotherapy)>
  > Pemetrexed: Dose frequency of Q3W, Day 1 of each cycle (standard Chemotherapy)
- Arm B Squamous Carcinoma (Pembro, Then MK-3475, Then Platinum Doublet, Then Maintenance MK-3475): For Squamous Carcinoma:> > Carboplatin AUC = 6 IV day 1 every 21-days for up to 4 cycles>
  > Paclitaxel 200 mg/m2 IV day 1 every 21-days for up to 4 cycles>
  > Carboplatin: Dose frequency of Q3W, Day 1 of each cycle (standard Chemotherapy)>
  >
  > Paclitaxel: Dose frequency of Q3W, Day 1 of each cycle (standard Chemotherapy)>
  > Pemetrexed: Dose frequency of Q3W, Day 1 of each cycle (standard Chemotherapy)
- Arm B Non-squamous Carcinoma (Pembro, Then MK-3475, Then Platinum Doublet, Then Maintenance MK-3475): For Non-squamous Carcinoma> > Carboplatin AUC = 6 IV day 1 every 21-days for up to 4 cycles>
  > Pemetrexed 500 mg/m2 IV day 1 every 21-days for up to 4 cycles>
  > MK-3475: Dose frequency of Q3W, Day 1 of each cycle>
  > Carboplatin: Dose frequency of Q3W, Day 1 of each cycle (standard Chemotherapy)>
  > Paclitaxel: Dose frequency of Q3W, Day 1 of each cycle (standard Chemotherapy)>
  > Pemetrexed: Dose frequency of Q3W, Day 1 of each cycle (standard Chemotherapy)
Period: Arm B Pembro Lead in Phase
Arm/Group | Arm A Squamous Carcinoma (Platinum Doublet, Then MK-3475, Then Maintenance MK-3475) | Arm A Non-squamous Carcinoma (Platinum Doublet, Then MK-3475, Then Maintenance MK-3475) | Arm B Squamous Carcinoma (Pembro, Then MK-3475, Then Platinum Doublet, Then Maintenance MK-3475) | Arm B Non-squamous Carcinoma (Pembro, Then MK-3475, Then Platinum Doublet, Then Maintenance MK-3475)
Started | 9 | 34 | 11 | 37
Completed | 9 | 34 | 10 | 37
Not Completed | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Period: Platinum Doublet Arm A, MK-3475 Arm B
Arm/Group | Arm A Squamous Carcinoma (Platinum Doublet, Then MK-3475, Then Maintenance MK-3475) | Arm A Non-squamous Carcinoma (Platinum Doublet, Then MK-3475, Then Maintenance MK-3475) | Arm B Squamous Carcinoma (Pembro, Then MK-3475, Then Platinum Doublet, Then Maintenance MK-3475) | Arm B Non-squamous Carcinoma (Pembro, Then MK-3475, Then Platinum Doublet, Then Maintenance MK-3475)
Started | 9 | 34 | 10 | 37
Completed | 4 | 25 | 6 | 20
Not Completed | 5 | 9 | 4 | 17
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — Adverse Event | 1 | 2 | 0 | 2
Not completed — Lack of Efficacy | 1 | 3 | 4 | 12
Not completed — Death | 1 | 2 | 0 | 2
Not completed — Deemed ineligible | 0 | 1 | 0 | 0
Not completed — Withdrew to hospice | 1 | 0 | 0 | 1
Not completed — Non compliance | 1 | 0 | 0 | 0
Period: MK-3475 Arm A, Platinum Doublet Arm B
Arm/Group | Arm A Squamous Carcinoma (Platinum Doublet, Then MK-3475, Then Maintenance MK-3475) | Arm A Non-squamous Carcinoma (Platinum Doublet, Then MK-3475, Then Maintenance MK-3475) | Arm B Squamous Carcinoma (Pembro, Then MK-3475, Then Platinum Doublet, Then Maintenance MK-3475) | Arm B Non-squamous Carcinoma (Pembro, Then MK-3475, Then Platinum Doublet, Then Maintenance MK-3475)
Started | 4 | 25 | 6 | 20
Completed | 2 | 17 | 4 | 18
Not Completed | 2 | 8 | 2 | 2
Not completed — Adverse Event | 0 | 2 | 0 | 1
Not completed — Lack of Efficacy | 2 | 6 | 0 | 0
Not completed — Death | 0 | 0 | 1 | 1
Not completed — Alternative Therapy | 0 | 0 | 1 | 0
Period: Maintenance MK-3475
Arm/Group | Arm A Squamous Carcinoma (Platinum Doublet, Then MK-3475, Then Maintenance MK-3475) | Arm A Non-squamous Carcinoma (Platinum Doublet, Then MK-3475, Then Maintenance MK-3475) | Arm B Squamous Carcinoma (Pembro, Then MK-3475, Then Platinum Doublet, Then Maintenance MK-3475) | Arm B Non-squamous Carcinoma (Pembro, Then MK-3475, Then Platinum Doublet, Then Maintenance MK-3475)
Started | 2 | 17 | 4 | 18
Completed | 0 | 3 | 1 | 7
Not Completed | 2 | 14 | 3 | 11
Not completed — Adverse Event | 0 | 3 | 1 | 2
Not completed — Lack of Efficacy | 0 | 9 | 0 | 8
Not completed — Death | 0 | 1 | 1 | 0
Not completed — Physician discretion | 0 | 0 | 1 | 0
Not completed — Withdrew to hospice | 0 | 1 | 0 | 0
Not completed — In active treatment | 2 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Arm A Squamous Carcinoma: For Squamous Carcinoma>
  > Carboplatin AUC = 6 IV day 1 every 21-days for up to 4 cycles>
  > Paclitaxel 200 mg/m2 IV day 1 every 21-days for up to 4 cycles>
  > Carboplatin: Dose frequency of Q3W, Day 1 of each cycle (standard Chemotherapy)>
  > Paclitaxel: Dose frequency of Q3W, Day 1 of each cycle (standard Chemotherapy)>
  > Pemetrexed: Dose frequency of Q3W, Day 1 of each cycle (standard Chemotherapy)
- Arm A Non-squamous Carcinoma: For Non-squamous Carcinoma> > Carboplatin AUC = 6 IV day 1 every 21-days for up to 4 cycles>
  > Pemetrexed 500 mg/m2 IV day 1 every 21-days for up to 4 cycles>
  > Carboplatin: Dose frequency of Q3W, Day 1 of each cycle (standard Chemotherapy)>
  >
  >> Paclitaxel: Dose frequency of Q3W, Day 1 of each cycle (standard Chemotherapy)>
  >>
  >
  >> Pemetrexed: Dose frequency of Q3W, Day 1 of each cycle (standard Chemotherapy)
- Arm B Squamous Carcinoma: For Squamous Carcinoma:>
  > Carboplatin AUC = 6 IV day 1 every 21-days for up to 4 cycles>
  > Paclitaxel 200 mg/m2 IV day 1 every 21-days for up to 4 cycles>
  > Carboplatin: Dose frequency of Q3W, Day 1 of each cycle (standard Chemotherapy)>
  > Paclitaxel: Dose frequency of Q3W, Day 1 of each cycle (standard Chemotherapy)>
  > Pemetrexed: Dose frequency of Q3W, Day 1 of each cycle (standard Chemotherapy)
- Arm B Non-squamous Carcinoma: For Non-squamous Carcinoma> > Carboplatin AUC = 6 IV day 1 every 21-days for up to 4 cycles>
  > Pemetrexed 500 mg/m2 IV day 1 every 21-days for up to 4 cycles>
  > MK-3475: Dose frequency of Q3W, Day 1 of each cycle>
  > Carboplatin: Dose frequency of Q3W, Day 1 of each cycle (standard Chemotherapy)>
  > Paclitaxel: Dose frequency of Q3W, Day 1 of each cycle (standard Chemotherapy)>
  > Pemetrexed: Dose frequency of Q3W, Day 1 of each cycle (standard Chemotherapy)
- Total: Total of all reporting groups
Arm/Group | Arm A Squamous Carcinoma | Arm A Non-squamous Carcinoma | Arm B Squamous Carcinoma | Arm B Non-squamous Carcinoma | Total
Number analyzed (Participants) | 9 | 34 | 11 | 37 | 91
Age, Continuous [Median (Full Range); unit: years] | 65 [50 to 77] | 69 [40 to 83] | 67 [48 to 71] | 68 [48 to 80] | 68 [40 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 17 | 4 | 20 | 43
  Male | 7 | 17 | 7 | 17 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 34 | 11 | 37 | 91
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1 | 0 | 2
  Black or African American | 3 | 1 | 1 | 3 | 8
  White | 5 | 33 | 9 | 32 | 79
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) Per RECIST 1.1
Description: The primary objective of this randomized phase II trial to determine the overall response rate (ORR per RECIST 1.1) in Chemotherapy naive patients with stage IV NSCLC after the administration of standard platinum-based chemotherapy before MK-3475 (arm A) and administration of MK-3475 administered before standard platinum-based chemotherapy (arm B). Overall Response (OR) = CR + PR.
Time Frame: 18 Months
Population: All patients that started treatment are included in analysis.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Groups:
- Arm A (Both Squamous and Non-Squamous): For Squamous Carcinoma Carboplatin AUC = 6 IV day 1 every 21-days for up to 4 cycles Paclitaxel 200 mg/m2 IV day 1 every 21-days for up to 4 cycles OR For Non-squamous Carcinoma> Carboplatin AUC = 6 IV day 1 every 21-days for up to 4 cycles Pemetrexed 500 mg/m2 IV day 1 every 21-days for up to 4 cycles Carboplatin: Dose frequency of Q3W, Day 1 of each cycle (standard Chemotherapy) Paclitaxel: Dose frequency of Q3W, Day 1 of each cycle (standard Chemotherapy) Pemetrexed: Dose frequency of Q3W, Day 1 of each cycle (standard Chemotherapy)
- Arm B (Both Squamous and Non-Squamous): MK-3475 200 mg/m2 IV every 21-days for up to 4 cycles> >>
  >
  >> Patients with CR, PR, or SD by irRC will then be treated with:>
  >>
  >
  >> For Squamous Carcinoma:>
  >>
  >
  >> Carboplatin AUC = 6 IV day 1 every 21-days for up to 4 cycles>
  >> Paclitaxel 200 mg/m2 IV day 1 every 21-days for up to 4 cycles>
  >>
  >
  >> OR>
  >>
  >
  >> For Non-squamous Carcinoma>
  >>
  >
  >> Carboplatin AUC = 6 IV day 1 every 21-days for up to 4 cycles>
  >> Pemetrexed 500 mg/m2 IV day 1 every 21-days for up to 4 cycles>
  >>
  >
  >> MK-3475: Dose frequency of Q3W, Day 1 of each cycle>
  >>
  >
  >> Carboplatin: Dose frequency of Q3W, Day 1 of each cycle (standard Chemotherapy)>
  >>
  >
  >> Paclitaxel: Dose frequency of Q3W, Day 1 of each cycle (standard Chemotherapy)>
  >>
  >
  >> Pemetrexed: Dose frequency of Q3W, Day 1 of each cycle (standard Chemotherapy)
Arm/Group | Arm A (Both Squamous and Non-Squamous) | Arm B (Both Squamous and Non-Squamous)
Number analyzed (Participants) | 43 | 47
proportion of participants | 0.395 [0.249 to 0.541] | 0.404 [0.264 to 0.545]
Statistical Analysis 1: Comparison: Arm A (Both Squamous and Non-Squamous) vs Arm B (Both Squamous and Non-Squamous); Test type: Superiority; p = 0.2176, Fisher Exact

2. Secondary Outcome: Compare Progression-Free Survival (PFS) Per RECIST 1.1
Description: To compare the progression-free survival (PFS) per RECIST 1.1 in previously untreated patients with advanced NSCLC treated with first line carboplatin-based chemotherapy followed by MK-3475 to patients treated with MK-3475 prior to first-line carboplatin-based chemotherapy.
Time Frame: 24 Months
Population: All patients that were treated were included in analysis.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Arm A (Both Squamous and Non-Squamous): For Squamous Carcinoma>> Carboplatin AUC = 6 IV day 1 every 21-days for up to 4 cycles>> Paclitaxel 200 mg/m2 IV day 1 every 21-days for up to 4 cycles>>
  >> OR>>
  >> For Non-squamous Carcinoma>> Carboplatin AUC = 6 IV day 1 every 21-days for up to 4 cycles>> Pemetrexed 500 mg/m2 IV day 1 every 21-days for up to 4 cycles>>
  >> Carboplatin: Dose frequency of Q3W, Day 1 of each cycle (standard Chemotherapy)>>
  >> Paclitaxel: Dose frequency of Q3W, Day 1 of each cycle (standard Chemotherapy)>>
  >> Pemetrexed: Dose frequency of Q3W, Day 1 of each cycle (standard Chemotherapy)
- Arm B (Both Squamous and Non-Squamous): MK-3475 200 mg/m2 IV every 21-days for up to 4 cycles>> >> Patients with CR, PR, or SD by irRC will then be treated with:>>
  >> For Squamous Carcinoma:>>
  >> Carboplatin AUC = 6 IV day 1 every 21-days for up to 4 cycles>> Paclitaxel 200 mg/m2 IV day 1 every 21-days for up to 4 cycles>>
  >> OR>>
  >> For Non-squamous Carcinoma>>
  >> Carboplatin AUC = 6 IV day 1 every 21-days for up to 4 cycles>> Pemetrexed 500 mg/m2 IV day 1 every 21-days for up to 4 cycles>>
  >> MK-3475: Dose frequency of Q3W, Day 1 of each cycle>>
  >> Carboplatin: Dose frequency of Q3W, Day 1 of each cycle (standard Chemotherapy)>>
  >> Paclitaxel: Dose frequency of Q3W, Day 1 of each cycle (standard Chemotherapy)>>
  >> Pemetrexed: Dose frequency of Q3W, Day 1 of each cycle (standard Chemotherapy)
Arm/Group | Arm A (Both Squamous and Non-Squamous) | Arm B (Both Squamous and Non-Squamous)
Number analyzed (Participants) | 43 | 47
Months | 5.8 [4.4 to 10.6] | 4.0 [2.1 to 10.3]
Statistical Analysis 1: Comparison: Arm A (Both Squamous and Non-Squamous) vs Arm B (Both Squamous and Non-Squamous); Test type: Superiority; p = 0.84, Log Rank; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.67 to 1.64]

3. Secondary Outcome: Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability)
Description: To characterize the adverse events related to MK-3475 by frequency, type and grade in patients with Chemotherapy naive advanced NSCLC based on the sequence of administration with first-line chemotherapy. A count of participants experiencing an adverse event is summarized here, the detailed summary is in the adverse events section of this report.
Time Frame: 24 Months
Measure: Number; unit: participants
Groups:
- Arm A Squamous Carcinoma; Arm A Non-squamous Carcinoma; Arm B Squamous Carcinoma; Arm B Non-squamous Carcinoma: Pemetrexed: Dose frequency of Q3W, Day 1 of each cycle (standard Chemotherapy)
Arm/Group | Arm A Squamous Carcinoma | Arm A Non-squamous Carcinoma | Arm B Squamous Carcinoma | Arm B Non-squamous Carcinoma
Number analyzed (Participants) | 9 | 34 | 10 | 37
participants | 9 | 34 | 10 | 37

4. Other Pre Specified Outcome: Evaluate the ORR Per irRC
Description: To evaluate the ORR per irRC of MK-3475 administered prior to or after treatment with first-line carboplatin-based chemotherapy in patients with previously untreated NSCLC.
Time Frame: 24 Months
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Evaluate PFS Per irRC
Description: To evaluate the PFS per irRC of previously untreated patients with advanced NSCLC who are treated with MK-3475 administered prior to or after first-line carboplatin-based chemotherapy.
Time Frame: 24 Months
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Evaluate Response Duration of MK-3475
Description: To evaluate the response duration of MK-3475 based on schedule of administration with standard platinum-based chemotherapy in patients with previously untreated advanced NSCLC.
Time Frame: 24 Months
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Evaluate the Overall Survival (OS)
Description: To evaluate the overall survival (OS) of patients with previously untreated advanced NSCLC who received MK-3475 administered prior to or after treatment with first line carboplatin-based chemotherapy.
Time Frame: 24 Months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 24 months
Description: The descriptions and grading scales found in the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4 will be utilized for AE reporting.
Groups:
- MK-3475: MK-3475 200 mg Q3W
- Carboplatin + Pemetrexed: For Non-squamous Carcinoma Carboplatin AUC = 6 IV day 1 every 21-days for up to 4 cycles Pemetrexed 500 mg/m2 IV day 1 every 21-days for up to 4 cycles Carboplatin: Dose frequency of Q3W, Day 1 of each cycle (standard Chemotherapy) Paclitaxel: Dose frequency of Q3W, Day 1 of each cycle (standard Chemotherapy) Pemetrexed: Dose frequency of Q3W, Day 1 of each cycle (standard Chemotherapy)
- "Carboplatin + Paclitaxel": Carcinoma Carboplatin AUC = 6 IV day 1 every 21-days for up to 4 cycles Pemetrexed 500 mg/m2 IV day 1 every 21-days for up to 4 cycles MK-3475: Dose frequency of Q3W, Day 1 of each cycle Carboplatin: Dose frequency of Q3W, Day 1 of each cycle (standard Chemotherapy) Paclitaxel: Dose frequency of Q3W, Day 1 of each cycle (standard Chemotherapy) Pemetrexed: Dose frequency of Q3W, Day 1 of each cycle (standard Chemotherapy)
Arm/Group | MK-3475 | Carboplatin + Pemetrexed | "Carboplatin + Paclitaxel"
All-Cause Mortality (participants affected / at risk) | 35/67 | 10/47 | 5/13
Serious Adverse Events (participants affected / at risk) | 17/67 | 6/47 | 4/13
Other Adverse Events (participants affected / at risk) | 66/67 | 46/47 | 12/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-3475 (N=67) | Carboplatin + Pemetrexed (N=47) | "Carboplatin + Paclitaxel" (N=13)
Blood and lymph sys disorders - Oth Spec (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Heart failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal, conn tissue - Oth spec (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Nervous system disorders - Oth spec (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 3 (3) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-3475 (N=67) | Carboplatin + Pemetrexed (N=47) | "Carboplatin + Paclitaxel" (N=13)
Anemia (Blood and lymphatic system disorders) | 29 (63) | 16 (22) | 3 (5)
Blood and lymph sys disorders - Oth Spec (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac disorders - Other, specify (Cardiac disorders) | 2 (3) | 0 (0) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Heart failure (Cardiac disorders) | 1 (3) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 3 (3) | 2 (2) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 2 (2) | 1 (1) | 1 (1)
Hypothyroidism (Endocrine disorders) | 9 (10) | 3 (3) | 0 (0)
Blurred vision (Eye disorders) | 3 (3) | 1 (1) | 1 (1)
Dry eye (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 3 (3) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Eyelid function disorder (Eye disorders) | 1 (2) | 1 (1) | 0 (0)
Floaters (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Watering eyes (Eye disorders) | 6 (6) | 4 (4) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 11 (16) | 3 (3) | 1 (1)
Bloating (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 29 (37) | 20 (21) | 6 (7)
Diarrhea (Gastrointestinal disorders) | 12 (22) | 6 (6) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (4) | 1 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 5 (7) | 4 (6) | 0 (0)
Nausea (Gastrointestinal disorders) | 27 (40) | 26 (34) | 4 (7)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 7 (9) | 5 (7) | 4 (4)
Chills (General disorders) | 2 (2) | 2 (2) | 0 (0)
Edema face (General disorders) | 1 (1) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 14 (26) | 6 (6) | 3 (4)
Fatigue (General disorders) | 45 (74) | 29 (39) | 8 (8)
Fever (General disorders) | 3 (3) | 1 (1) | 1 (1)
Flu like symptoms (General disorders) | 1 (1) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 4 (4) | 1 (1) | 0 (0)
Gen disord and admin site conds-Oth spec (General disorders) | 4 (5) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 1 (1) | 0 (0)
Localized edema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 2 (2) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 13 (16) | 2 (3) | 2 (3)
Pain (General disorders) | 13 (32) | 6 (7) | 3 (5)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
Allergic reaction (Immune system disorders) | 2 (3) | 0 (0) | 1 (1)
Immune system disorders - Other, specify (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gum infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 4 (5) | 0 (0) | 1 (1)
Mucosal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 3 (4) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 5 (5) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (4) | 2 (2) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 6 (6) | 1 (1) | 2 (2)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Inj, pois and proced complic - Oth spec (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Activated partial throm time prolonged (Investigations) | 1 (1) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 3 (4) | 3 (3) | 0 (0)
Alkaline phosphatase increased (Investigations) | 6 (7) | 4 (4) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 4 (12) | 2 (3) | 1 (1)
Cardiac troponin T increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 3 (7) | 0 (0) | 1 (1)
INR increased (Investigations) | 2 (2) | 0 (0) | 1 (1)
Investigations - Other, specify (Investigations) | 1 (1) | 1 (1) | 1 (1)
Lymphocyte count decreased (Investigations) | 7 (23) | 1 (2) | 2 (7)
Neutrophil count decreased (Investigations) | 5 (9) | 6 (7) | 1 (1)
Platelet count decreased (Investigations) | 5 (14) | 5 (8) | 2 (2)
Weight gain (Investigations) | 1 (4) | 0 (0) | 1 (3)
Weight loss (Investigations) | 8 (14) | 2 (2) | 2 (2)
White blood cell decreased (Investigations) | 5 (8) | 6 (7) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 30 (39) | 16 (18) | 8 (8)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 9 (12) | 6 (6) | 3 (5)
Hyperkalemia (Metabolism and nutrition disorders) | 3 (4) | 1 (1) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 5 (12) | 0 (0) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 (13) | 2 (2) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 7 (9) | 5 (5) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 4 (6) | 0 (0) | 5 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 (21) | 5 (6) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (4) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (10) | 6 (6) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 2 (2) | 0 (0)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 6 (6) | 3 (3) | 2 (2)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 1 (1)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Musculoskeletal, conn tissue - Oth spec (Musculoskeletal and connective tissue disorders) | 5 (6) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 9 (9) | 2 (2) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 (17) | 5 (7) | 1 (1)
Ataxia (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Concentration impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 10 (11) | 7 (8) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 14 (15) | 7 (7) | 2 (3)
Facial muscle weakness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 13 (19) | 2 (2) | 1 (1)
Lethargy (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 13 (18) | 6 (7) | 6 (6)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 3 (3) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 11 (16) | 5 (5) | 1 (2)
Depression (Psychiatric disorders) | 12 (12) | 5 (5) | 2 (2)
Insomnia (Psychiatric disorders) | 21 (25) | 11 (13) | 3 (3)
Libido decreased (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 3 (3) | 0 (0) | 0 (0)
Renal and urinary disorders - Oth spec (Renal and urinary disorders) | 2 (3) | 1 (2) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 3 (3) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 1 (1) | 2 (2) | 0 (0)
Urinary urgency (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0)
Penile pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 31 (35) | 15 (15) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 27 (40) | 14 (17) | 5 (7)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 3 (3) | 1 (1)
Pharyngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 2 (2) | 2 (2)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2) | 1 (1)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 7 (12) | 5 (5) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 10 (12) | 3 (3) | 4 (4)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Nail discoloration (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Nail ridging (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 17 (19) | 5 (5) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 14 (18) | 7 (8) | 3 (4)
Scalp pain (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 7 (10) | 1 (1) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 0 (0)
Surgical and medical proced - Oth spec (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Hot flashes (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 9 (17) | 4 (5) | 2 (4)
Hypotension (Vascular disorders) | 1 (2) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-14): https://cdn.clinicaltrials.gov/large-docs/15/NCT02591615/Prot_SAP_000.pdf